CLINICAL TRIAL: NCT02240043
Title: Growth Hormone Evaluation in the Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Ana Beatriz Winter Tavares, MD, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 185/09; Memo n 019/10 (Registry Identifier: Comite de ética e Pesquisa HUCFF)
Record Dates: First submitted 2014-08-31; First posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- growth hormone secretion (Other): The elderly had common morbidities peculiar to their age, such as systemic arterial hypertension, diabetes mellitus, Parkinson's disease, initial stages of senile dementia, and osteoporosis.
  Interventions: Other: growth hormone secretion

INTERVENTIONS:
Other: growth hormone secretion — The glucagon stimulation test (GST) was performed by intramuscular injection of 1 mg of glucagon (Glucagen® Hypokit, Novo Nordisk A/S, Denmark). The blood samples were collected at baseline and after 90 minutes, 120 minutes, 150 minutes and 180 minutes of glucagon injection for GH and cortisol measurements. The subjects were recumbent during the test, and a cannula was maintained in a vein in the arm or forearm with a saline solution slowly infused to avoid multiple punctures.

SUMMARY:
The aim of this study is to evaluate the growth hormone (GH) and adrenocorticotrophic hormone (ACTH) secretion in elderly without hypothalamic-pituitary disease using the glucagon stimulation test (using Glucagen® Hypokit, Novo Nordisk A/S, Denmark) and evaluate some parameters such as sarcopenia, nutritional state, bone mineral density, frailty criteria with secretion of GH.

DETAILED DESCRIPTION:
subjects over 65 years old were recruited from the geriatric ambulatory unit of our hospital to voluntarily participate in a research study concerning the GH and ACTH axis in the elderly, which included the realization of the glucagon stimulation test as the first phase of the study.

The GST (Glucagen® Hypokit, Novo Nordisk A/S, Denmark) was the chosen test to assess both ACTH and GH release because of its few known contraindications and mild side effects. It is a provocative test to evaluate GH and ACTH axis, i.e, a diagnostic test, without therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* elderly people above 65 years old with comorbidities peculiar to their age (such as hypertension, diabetes, dyslipidemia, parkinson disease) or without comorbidities

Exclusion Criteria:

* pituitary disease, severe acute disease, terminal renal chronic disease, active malignant cancer, the presence of any other disease that could interfere with the somatotrophic axis evaluation, and the contraindications for glucagon administration (pheochromocytoma, insulinoma and malnourishment).

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Growth Hormone Secretion in the elderly people using glucagon stimulation test (GST) | up to one week

SECONDARY OUTCOMES:
ACTH release in the elderly people using GST | up to one week
  ACTH: adrenocorticotrophic hormone

OTHER OUTCOMES:
Body composition in the elderly people according with GH secretion | up to 3 months
  To realize Dual-energy X-ray absorptiometry (DEXA) to evaluate body composition after the realization of the Glucagon stimulation test. It could take some time to be done because of availability of the equipment

CONTACTS AND LOCATIONS:
Overall Officials: Flávia L Conceição, PhD, Study Director — Hospital Universitário Clementino Fraga Filho - UFRJ

REFERENCES:
- [Derived] Tavares AB, Seixas-da-Silva IA, Silvestre DH, Paixao CM Jr, Vaisman M, Conceicao FL. Potential risks of glucagon stimulation test in elderly people. Growth Horm IGF Res. 2015 Feb;25(1):53-6. doi: 10.1016/j.ghir.2014.11.002. Epub 2014 Nov 29. PMID 25481820